CLINICAL TRIAL: NCT03613948
Title: Study on the Effects of Mutations Under Inherited Retinal Disease in Korean
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jinu Han, Associate Professor, Gangnam Severance Hospital
Other Study IDs: 3-2018-0026
Record Dates: First submitted 2018-04-10; First posted 2018-08-03 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Inherited Retinal Dystrophy Primarily Involving Sensory Retina; Inherited Retinal Dystrophy Primarily Involving Retinal Pigment Epithelium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood DNA samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop comprehensive genetic maps of inherited retinal diseases in Korean

* Establishment of comprehensive genetic database in Koreans with inherited retinal diseases including frequently mutated genes, genotype-phenotype correlations, and visual prognosis."

DETAILED DESCRIPTION:
Group/ Cohort Label : Subject with age between 6 months and 65 years who have not receive molecular genetic testing Group / Cohort Description : Consecutive subjects with inherited retinal disease who are willing to do genetic testing using whole exome sequencing (n=265) and whole genome sequencing (n=15) and agree to informed consent of the study

ELIGIBILITY:
Inclusion Criteria:

* Inherited retinal disease
* Age between 4 months and 75 years
* Subject who has clinically confirmed visual impairment including night blindness or photophobia. Subject should meet one of the following criteria
* pigmentary retinopathy in both eyes
* reduced response in photopic or scotopic electroretinogram in both eyes
* photoreceptor degeneration in optical coherence tomography in both eyes

Exclusion Criteria:

* unilateral retinal disease
* Subject who had previously confirmed genetic testing
* Age less than 4 months or more than 75 years
* When congenital infection or trauma are suspicious for the cause of retinal disease
* When age-related macular degeneration, myopic degeneration, autoimmune origin are suspicious for the cause of retinal disease
* No visual impairment or normal electroretinogram (e.g., benign fleck)
* Illiterate subject who can not understand informed consent
* Foreigners

Ages: 4 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: "Subject with inherited retinal disease, age between 6 months and 75 years who have not receive molecular genetic testing"
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic rate of whole exome sequencing (n=265) in Koreans with inherited retinal disease | 3 years (until December 31, 2020)
  patients were grouped in 1) probable molecular diagnosis: patients with pathogenic or likely pathogenic disease-associated variant(s), 2) possible molecular diagnosis: patients with 2 heterozygous mutations without segregation analysis, or patients harboring a single pathogenic or likely pathogenic disease-associated variant in a gene linked with recessive traits, provided the patient phenotype matches the known spectrum of clinical features for this gene, 3) unsolved: all other patients for which no pathogenic or likely pathogenic disease-associated variants were detected.

SECONDARY OUTCOMES:
Diagnostic rate of whole genome sequencing (n=15) in Koreans with inherited retinal disease | 3 years (until December 31, 2020)
  patients were grouped in 1) probable molecular diagnosis: patients with pathogenic or likely pathogenic disease-associated variant(s), 2) possible molecular diagnosis: patients with 2 heterozygous mutations without segregation analysis, or patients harboring a single pathogenic or likely pathogenic disease-associated variant in a gene linked with recessive traits, provided the patient phenotype matches the known spectrum of clinical features for this gene, 3) unsolved: all other patients for which no pathogenic or likely pathogenic disease-associated variants were detected.

CONTACTS AND LOCATIONS:
Overall Officials: Jinu Han, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Result] Stone EM, Andorf JL, Whitmore SS, DeLuca AP, Giacalone JC, Streb LM, Braun TA, Mullins RF, Scheetz TE, Sheffield VC, Tucker BA. Clinically Focused Molecular Investigation of 1000 Consecutive Families with Inherited Retinal Disease. Ophthalmology. 2017 Sep;124(9):1314-1331. doi: 10.1016/j.ophtha.2017.04.008. Epub 2017 May 27. PMID 28559085